CLINICAL TRIAL: NCT02772952
Title: Effectiveness of a Multi-componentphysical Training Integrated Into a Multimodal Program Based on the Evidence in Hiper-fragile Elders: A Randomized Clinical Trial STUDY POWER_AGING
Brief Title: Effectiveness of a Multi-component Physical Training in Hyper-fragile Elders: A Randomized Clinical Trial
Acronym: PowerA-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Collaborators: Andaluz Health Service (Other Government)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, Professor, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Power-Aging-01
Record Dates: First submitted 2015-12-02; First posted 2016-05-16 (Estimated); Last update posted 2024-06-04 (Actual); Status verified 2019-05

CONDITIONS: Multimodal Intervention; Fragility; Other Metabolic Diseases; Physical Activity; Patient Fall; Dietary Modification
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): a control group whose intervention will be to review medication + adequacy of diet + health education (physical activity recommendation (within a comprehensive advice on healthy lifestyles)
  Interventions: Other: Control Intervention
- Experimental Group (Experimental): Experimental group whose intervention will be a Multimodal Intervention: therapeutic exercise + review medication + adequacy of diet + health education program.
  Interventions: Other: Multimodal Intervention

INTERVENTIONS:
Other: Control Intervention — Control Intervention: review medication + adequacy of diet + health education (physical activity recommendation (within a comprehensive advice on healthy lifestyles)
  Arms: Control Group
Other: Multimodal Intervention — Multimodal Intervention: therapeutic exercise + review medication + adequacy of diet + health education program
  Arms: Experimental Group

SUMMARY:
Objective: To compare short-term and medium-term effectiveness of a multimodal program that integrates a program of therapeutic exercise, medication review, adequacy of diet and health education, compared with standard medical practice in improving neuromuscular and physiological status on frail elderly. Another aim is to analyze the maintenance of these effects by monitoring long-term (12 months) from the start of the intervention.

Design: Randomized controlled trial Scope / Study subjects: recruited frail elderly in Basic Health Zone of Malaga. Methods: The subjects to be included in the study (after meeting inclusion / exclusion) will be randomized into two groups: a control group whose intervention will be to review medication + adequacy of diet + health education (physical activity recommendation (within a comprehensive advice on healthy lifestyles) and an experimental group whose intervention will be a Multimodal Intervention: therapeutic exercise + review medication + adequacy of diet + health education program.

Sociodemographic, Clinical and monitoring Variables will be collected at baseline. Moreover, tracking variables will be collected at 2 and 6 months after starting the intervention and at 3 and 6 months after the end of the intervention (monitoring).

The monitoring variables that will be measured are: BMI , general health, fatigue, brittleness, Motor Control, Attention - Concentration - Memory, Motor Memory , spatial orientation, grip strength, balance (static - semi-static and dynamic ), gait speed and metabolomic variables.

One descriptive analysis of the sociodemographic variables of the participants will be performed. Further the change on the variables intra-subjects (pre-post intervention) and inter-subjects (experimental group vs control group) will be calculated. For the intra-subject analysis will be performed a ANOVA-one factor analysis. The intersubject outcome variables will be compared between the two groups in each moments of data collection, using the student t-test or Wilconxon (depending of the sample distribution). The level of significance was set at P ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* People 65 years older than after screening of fragility as the test battery Short Physical Performance Battery (SPPB), can perform the therapeutic exercise program

Exclusion Criteria:

* Presence in the medical history of neuromuscular , metabolic, hormonal and / or cardiovascular disorders.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 114 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Body mass index | Baseline - 6 months after the end of the intervention
  The measurements will be taken following the anthropometric parameter guidelines of The International Society for the Advancement of Kinanthropometry (ISAK) (Ross et al., 1978).
Health Related Quality of Life SF-12 | Baseline - 6 months after the end of the intervention
  General health condition was measured using the SF-12 short form questionnaire, adapted from the extended SF-36 version. Both physical and mental components are evaluated. The higher the score the better the condition. SF-12 reliability has proven a high internal consistency demonstrating an approximate ICC (Intraclass Correlation Coefficient) of 0.9. (Vigalut et al., 2008).
Fatigue State POMS (Profile of Mood States) | Baseline - 6 months after the end of the intervention
  The Spanish version of POMS published by Andrade et al. (2010) was used, with 44 items that represented six conceptual dimensions: anger (11 items), fatigue (6 items), vigour (5 items), friendship (6 items), stress (7 items) and depressed state (9 items). As usual, the answer format consisted of a 5 ordered category response, assigned with values 0 (nothing) to 4 (a lot). All the items were put forward in the same trend except for the item 29-relaxed (corresponding to the state of stress) scores, that were inverted after the test.
Frailty Questionnaire | Baseline - 6 months after the end of the intervention
  The auto-administrated survey based in 10 dichotomous questions in order to detect elder frail people will be carried out (Di Bari et al.2014).
MMSE (Mini-Mental State Examination) - MEC-30 (Mini Cognitive Examination | Baseline - 6 months after the end of the intervention
  The MEC consists of 30 items grouped into 11 sections (Fig. 1), the clinician could carry out in 5-15 min based on the following indications; note that those responsible for carrying out this instrument, both in its original version (Folstein) and its Spanish adaptation (Lobo et al, 2002), warn that the professional should stick to these criteria as far as possible, ensuring maximum objectivity in registering the subject's responses. The eleven sections are: Orientation to time, Orientation to space, Registration, Attention and Calculation, Memory, Nomination, Repetition (Recall), Comprehension, Reading, Writing and Drawing.
Motor memory test | Baseline - 6 months after the end of the intervention
  Motor skill memory and body awareness will be measured directing a test that consists of performing ten static positions. The examiner executes 10 positions holding each one of them for 10 seconds. Immediately after, the patient imitates the position in the opposite way, analogous to a mirror. The test ends when the 10 positions have been carried out. This test is included in the "Memory in movement" program, used as a cognitive intervention tool (Rey Cao, Canales Lacruz, Táboas País, & Cancela Carra, 2008).
Spatial orientation test | Baseline - 6 months after the end of the intervention
  The SODT-R (Spatial Orientation Dynamic Test-Revised, SODT-R, Colom, Contreras, Shih and Santacreu, 2003) task is to direct two moving objects to a given destination. There are two buttons for each of the moving objects in order to control their course, as shown in Figure 1. Pressing the buttons changes the object's course in one direction, reducing or increasing the angular discrepancy between the current course compared to the ideal course that would stand for 0 deviation.
Grip strength test | Baseline - 6 months after the end of the intervention
  Hand grip strength test will examine the peak of strength and fatigue resistance. The test is performed with the participant in a sitting position and 90 degree elbow flexion, neutral pronosupination and flexion, extension or inclination of the wrist will not be allowed. The patient will be asked to hand grip, which will be evaluated with a hydraulic dynamometer JAMAR (Bellace, Healy, Besser, Byron, & Hohman, 2000).
Balance (static - semi-static and dynamic) test | Baseline - 6 months after the end of the intervention
  Expanded TUG is a test to assess mobility, balance and risk of falls in the elderly. (Podsiadlo and Richardson, 2015). The test consists of timing how long the seated patient takes to get up, walk ten metres, return and sit back again on the chair.

CONTACTS AND LOCATIONS:
Locations (1):
- Antonio Cuesta-Vargas, Málaga, Spain

REFERENCES:
- [Derived] Gonzalez-Sanchez M, Cuesta-Vargas AI, Del Mar Rodriguez Gonzalez M, Caro ED, Nunez GO, Galan-Mercant A, Belmonte JJB. Effectiveness of a muticomponent workout program integrated in an evidence based multimodal program in hyperfrail elderly patients: POWERAGING randomized clinical trial protocol. BMC Geriatr. 2019 Jun 21;19(1):171. doi: 10.1186/s12877-019-1188-x. PMID 31226936